CLINICAL TRIAL: NCT03946592
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Phase Ⅲ Clinical Trial to Evaluate the Efficacy and Safety of DWJ211 in Patient With Moderate or Severe Submental Fat
Brief Title: Evaluate the Efficacy and Safety of DWJ211 in Patient With Moderate or Severe Submental Fat
Acronym: SMF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DW_DWJ211301
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Submental Fat
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Inject the Drug into submental fat via subcutaneous
  Interventions: Drug: Normal saline
- DWJ211 group (Experimental): Inject the Drug into submental fat via subcutaneous
  Interventions: Drug: DWJ211

INTERVENTIONS:
Drug: Normal saline — Inject the Drug into submental fat via subcutaneous
  Arms: Placebo group
Drug: DWJ211 — Inject the Drug into submental fat via subcutaneous
  Arms: DWJ211 group

SUMMARY:
Evaluate the efficacy and safety of DWJ211 in patient with moderate or severe submental fat

DETAILED DESCRIPTION:
DWJ211 is a injectable drug for improvement in the appearance of moderate to severe submental fat (SMF)

ELIGIBILITY:
Inclusion Criteria:

* Submental fat grade by the investigator as 2 or 3 using the PA-SMFRS and graded by the subject as 2 or 3 using the SA-SMFRS as determined on Visit 1.
* Dissatisfaction with the submental area expressed by the subject as a rating of 1~3 using the SSS as determinded on Visit 1.
* Less than 35kg/m2 in body mass index on Visit1.
* Subject who will agree with the no treatment for the procedure that may affect to reduction or the submental fat.

Exclusion Criteria:

* History of any intervention to treat SMF
* History of trauma associated with the chin or neck areas that in the judgement of the investigator may affect evaluation of safety or efficacy of treatment.
* Evidence of any cause of enlargement in the submental area.
* History or current symptoms of dysphagia.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
PA-SMFRS, SA-SMFRS | 12 week after last treatment
  Proportion of subject who simultaneously have at least a 1 grade, 2grade improvement from baseline on the PA-SMFRS, SA-SMFRS after the last treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-ang university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No